CLINICAL TRIAL: NCT04686838
Title: READyR-II: Dynamic Tailoring Phase for a Remote Assessment and Dynamic Response Intervention to Support Couples in Planning for Changing Dementia Care Needs
Brief Title: REmote Assessment and Dynamic Response Intervention II
Acronym: READyR-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lyndsey Miller, Co-Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-2; P30AG024978-17 (NIH)
Record Dates: First submitted 2020-12-16; First posted 2020-12-29 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Dementia; Alzheimer Disease; Relationship, Marital; Caregiver Stress Syndrome
Keywords: Needs Assessment; Remote Monitoring; Technology; Care Values; Aging-in-Place; Family Caregiver
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Dyads will be randomized (assigned by chance) to one of two groups: 1) READyR A or 2) READyR B
Who Masked: Participant
Masking Description: Participants will all agree to the dynamic tailoring phase with remote monitoring and surveys, and will not know whether the phone calls are related to anomaly detection or are a control condition phone call.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- READyR II A (Experimental): Continuous monitoring will be conducted and analyzed for anomaly detection. Participants in this arm will receive contact phone call when a potential change in care needs is indicated by an anomaly.
  Interventions: Behavioral: READyR II: A
- READyR II B (comparison) (Active Comparator): Sensors will remain in the home but anomaly detection analysis will not be performed and contact phone calls will be at regular intervals without dynamic tailoring content. Standard educational content will instead be shared over the phone.
  Interventions: Behavioral: READyR II: B

INTERVENTIONS:
Behavioral: READyR II: A — Continuous monitoring for anomaly detection and contact phone call when a potential change in care needs is indicated by an anomaly.
  Arms: READyR II A
Behavioral: READyR II: B — Sensors will remain in the home but anomaly detection analysis will not be performed and contact phone calls will be at regular intervals without dynamic tailoring content.
  Arms: READyR II B (comparison)

SUMMARY:
The purpose of the READyR II Study is to test a dynamic tailoring phase of a remote assessment for changing dementia-related care needs.

DETAILED DESCRIPTION:
Unmet dementia-related care needs are highly prevalent, and are detrimental to the care dyad's (person with dementia and their family care partner) health, safety, mortality, and likelihood of nursing home placement. READyR II tests a dynamic tailoring phase of an intervention program that was previously developed to remotely assess dementia-related care needs using digital data on behavioral patterns (from sensors and wearables) in the home. READyR II follows participants who have completed READyR for a total of six months in order to detect anomalies in activity patterns that may indicate new and unforeseen care needs.

People who voluntarily decide to participate in this follow-up intervention study will be asked to continue participating with the in-home monitoring sensor platform, complete weekly questionnaires, and receive regular follow-up telephone calls from the study team.

ELIGIBILITY:
Inclusion Criteria:

* 62 years or older;
* Able to identify a family care partner over age 20 who is living with you and will also consent to fully participate in the study
* Probable or confirmed diagnosis of mild cognitive impairment or early-stage dementia
* Age and education adjusted MOCA score > 15 (at most recent measurement by parent study) corresponding to early to moderate stage dementia

Exclusion Criteria:

* Inability to speak English or read printed materials in English
* Conditions that would limit participation at entry to study (e.g. visual or hearing impairments prohibiting reading and discussing the intervention materials)
* Any uncontrolled medical condition that is expected to preclude completion of the study, such as late stage cancers

Family Care Partners

Inclusion:

* 21 years or older;
* Self-identifying as a family member and care partner residing with the PwD participant;

Exclusion:

* Inability to speak English or read printed materials in English
* Conditions that would limit participation at entry to study (e.g. visual or hearing impairments prohibiting reading and discussing the intervention materials);
* Any uncontrolled medical condition that is expected to preclude completion of the study, such as late stage cancers.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Mean difference effect sizes for pre-post change the care dyad's preparation for future care needs | Baseline compared with 18 weeks
  The Preparation for Future Care Needs Scale (Short Form) assesses the degree to which an individual has engaged in planning for future care needs in late life using 15 items and 5 subscales representing distinct planning processes (awareness, gathering information, decision making, concrete planning, avoidance). Items are scored on a 5 point Likert scale with higher scores indicating greater preparation for future care needs.
  Sorensen, S., Chapman, B. P., Duberstein, P. R., Pinquart, M., & Lyness, J. M. (2017). Assessing future care preparation in late life: Two short measures. Psychol Assess, 29(12), 1480-1495.
Mean difference effect sizes for pre-post change in the care dyad's relationship quality | Baseline compared with 18 weeks
  The Dyadic Relationship Scale assesses the positive dyadic interactions and negative dyadic strain experienced by caregivers (11 items) and care recipients (10 items). Items are averaged for a summary score that ranges from 0 to 3, with higher scores indicating more positive interactions in the relationship, or more relationship strain, respectively.
  Sebern, M.D. & Whitlatch, C.J. (2007). Dyadic Relationship Scale: A measure of the impact of the provision and receipt of family care. The Gerontologist, 47(6), 741-751.
Mean difference effect sizes for pre-post change in the amount of incongruence between the care partner's understanding of the care values of the person with dementia | Baseline compared with 18 weeks
  The Care Values Scale assesses the importance of four care-related values to the person with dementia from the perspectives of the person with dementia and their care partner. Items for each of the four subscales are averaged for a summary score that ranges from 1 to 3, with higher scores indicating greater importance of the care value to the person with dementia.
  Miller LM, Whitlatch CJ, Lee CS, Caserta MS. Care Values in Dementia: Patterns of Perception and Incongruence Among Family Care Dyads. The Gerontologist. 2018.

SECONDARY OUTCOMES:
Mean difference effect sizes for pre-post change in the amount of care-related strain reported | Baseline compared with 12 weeks
  Subjective strain from caregiving will be assessed among family care partners at baseline and follow-up assessments using the Zarit Burden Interview (ZBI), short-form (12 items). Scores range from 0-48 with higher scores indicating a greater degree of strain from providing care.
Mean difference effect sizes for pre-post change in the care dyad's quality of life | Baseline compared with 18 weeks
  The Quality of Life: Alzheimer's Disease Scale assesses individual perceptions of quality of life (from poor to excellent) across 13 items. Items are averaged for a summary score of 1 to 4, higher scores indicating greater degree of quality of life. Logsdon, R. G., Gibbons, L. E., McCurry, S. M., & Teri, L. (1999). Quality of Life in Alzheimer's Disease: Patient and Caregiver Reports. Journal of Mental Health and Aging, 5(1), 21-32.
Mean difference effect sizes for pre-post change in the care dyad's concealment of emotions | Baseline compared with 18 weeks
  The Emotional Intimacy Disruptive Behavior Scale (8 items) assesses the frequency of engagement in behaviors to conceal emotions about an illness from one's partner. Druley, J. A., Stephens, M. A. P., & Coyne, J. C. (1997). Emotional and physical intimacy in coping with Lupus: Women's dilemmas of disclosure and approach. Health Psychology, 16, 506-514.

OTHER OUTCOMES:
Time spent out of the home | Continuously over 18 weeks
  Time spent out of home will be robustly and accurately measured through an algorithm using sensor (motion/contact) and actigraphy data.
  Petersen J, Austin D, Mattek N, Kaye J. Time Out-of-Home and Cognitive, Physical, and Emotional Wellbeing of Older Adults: A Longitudinal Mixed Effects Model. PloS one. 2015;10(10):e0139643.
Physical activity / sedentary behavior | Continuously over 18 weeks
  Physical activity and sedentary bouts will be measured using actigraphy data.
Time spent together / separate | Continuously over 18 weeks
  Time spent together/separate as a dyad will be observed through previously-developed algorithms using data from PIR motion/contact sensors and actigraphy. We will consider times when the informal care dyad is together in the same room, separate within/outside of the home, and time in bathroom together (indicating ADL dependency).
Sleep patterns | Continuously over 18 weeks
  Sleep patterns be measured using actigraphy, motion sensors, and a bed mat sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Lyndsey M Miller, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be available upon request to our Alzheimer's Disease Research Center
  Supporting Information:
  Time Frame:
  Data will become available after completion of study and after publication of primary study aims.
  Access Criteria:
  Requests need to made to the PI at the Oregon Alzheimer's Disease Research Center (OARDC). A short data request form will need to be submitted to the OADRC.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code